CLINICAL TRIAL: NCT03010306
Title: Pilot Community-based Development Intervention (CASITA) for Children With Neurodevelopmental Risk and Delay in Carabayllo, Lima, Peru
Brief Title: CASITA Intervention for Children at Risk of Delay in Carabayllo, Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Grand Challenges Canada (Other); Harvard University (Other); Boston Children's Hospital (Other); Boston Medical Center (Other); Partners in Health (Other)
Responsible Party: Principal Investigator, Adrianne Katrina Hart Nelson, Research Manager, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002554
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Child Developmental Delay; Child Development; Community Health Workers; Low Income Population
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition only (No Intervention): Monthly food baskets were provided to the nutrition only group. Food baskets included basic foods to sustain a family of three over one month's time, such as rice and evaporated milk. Food baskets were valued at approximately $28 US Dollars per basket.
- Nutrition + CASITA (Active Comparator): The CASITA intervention was given by a community health worker (CHW) and involves individual and group modalities. HOME-CASITA took place at the dyad's place of residence, and the GROUP-CASITA at a local community center. All CASITA participants received 12 weekly sessions over 3 months. Interventions retain core elements of the SPARK approach: coaching parents on child development stimulation and providing social support and encouragement. Each session is as follows: 1) Child observation & knowledge sharing about child development; 2) Practice of reciprocal attention focusing and social interaction activities; 3) Parent encouragement on behavior and developmental interactions; and 4) Parent social support through referral assistance, reassurance, and validation of parent's concerns.
  Interventions: Other: CASITA

INTERVENTIONS:
Other: CASITA
  Other Names: Child development coaching and social support in Lima Peru; Community-based intervention for children at risk of Neurodevelopment delay
  Arms: Nutrition + CASITA

SUMMARY:
Building on an intervention for early child development from the SPARK Center in Boston, Socios En Salud (SES) pilot tested "CASITA" a community-based package to screen and treat young children (ages 1-3 years of age) diagnosed with neurodevelopment risk and delay in Carabayllo, Lima, Peru. Ministry of Health CHWs identified children with developmental delays within the clinics and community and delivered a structured early intervention that included parent coaching and social support. In order to test the hypothesis that CASITA improves early child development, caregiver, and home environment, dyads received either nutrition supplements alone, nutrition + "CASITA" early child development sessions individually, or CASITA in a group of 10 dyads.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 - 24 months of age;
2. Known primary caregiver (parent or legal guardian) living with child;
3. Living within the catchment area of the 6 Health Centers that comprise the study zone.
4. Screen positive for neurodevelopment delay ("at risk" or "delayed" in neurodevelopment based on Evaluation del Desarrollo Psicomotor (EEDP) assessment).
5. Be at risk by scoring <45 on the Progress Out of Poverty Index.

Exclusion Criteria:

1. A known medical condition that would make the child unresponsive to early intervention;
2. Family anticipates moving within the next three months.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in risk of delay, as measured by the EASQ | baseline, 3 months
  The Ages and Stages Questionnaire (ASQ) is an internationally-validated instrument that can be used to assess change in developmental risk over time. Fernald et al incorporated additional observation-based assessments and the following modifications: 1) addition of child observation exercises to allow for validity check of parent responses (original ASQ questions), and 2) the incorporation of ASQ questions from the next highest age range. The Extended Ages and Stages Questionnaire (EASQ) was utilized as an assessment tool to allow us to better quantify degree of risk at baseline (based on quintiles of scores). By incorporating ASQ questions from the next two highest age ranges, scores will be continuous across the study period of three. The EASQ has been applied to children in four countries, including 2,845 children in Peru.

SECONDARY OUTCOMES:
Change in global HOME score | baseline, 3 months
  The Infant Toddler Home Observation Measurement of the Environment (HOME) evaluates parenting and home influences on child development.
Change in HOME subscore of parent responsivity | baseline, 3 months
  This HOME subscore is defined in the manual as "the extent to which the parent responds to the child's behavior including reinforcement for desired behavior and communication through words and actions".
Change in HOME subscore of parent involvement | baseline, 3 months
  This HOME subscore is defined as "parental acceptance of the child's behavior that is less than optimal and examines avoidance of undue restriction and punishment".

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Lecca, MD, Principal Investigator — Socios En Salud, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grantham-McGregor S, Cheung YB, Cueto S, Glewwe P, Richter L, Strupp B; International Child Development Steering Group. Developmental potential in the first 5 years for children in developing countries. Lancet. 2007 Jan 6;369(9555):60-70. doi: 10.1016/S0140-6736(07)60032-4. PMID 17208643
- [Background] Nahar B, Hamadani JD, Ahmed T, Tofail F, Rahman A, Huda SN, Grantham-McGregor SM. Effects of psychosocial stimulation on growth and development of severely malnourished children in a nutrition unit in Bangladesh. Eur J Clin Nutr. 2009 Jun;63(6):725-31. doi: 10.1038/ejcn.2008.44. Epub 2008 Sep 3. PMID 18772893
- [Background] Nahar B, Hossain MI, Hamadani JD, Ahmed T, Huda SN, Grantham-McGregor SM, Persson LA. Effects of a community-based approach of food and psychosocial stimulation on growth and development of severely malnourished children in Bangladesh: a randomised trial. Eur J Clin Nutr. 2012 Jun;66(6):701-9. doi: 10.1038/ejcn.2012.13. Epub 2012 Feb 22. PMID 22353925
- [Background] Munoz M, Bayona J, Sanchez E, Arevalo J, Sebastian JL, Arteaga F, Guerra D, Zeladita J, Espiritu B, Wong M, Caldas A, Shin S. Matching social support to individual needs: a community-based intervention to improve HIV treatment adherence in a resource-poor setting. AIDS Behav. 2011 Oct;15(7):1454-64. doi: 10.1007/s10461-010-9697-9. PMID 20383572
- [Background] Caldwell, B. and R. Bradley, eds. Home Inventory Administration Manual. 3rd Edition ed. 2001, University of Arkansas at Little Rock: Little Rock, AR.
- [Background] Schreiner, M., Progress out of Poverty Index: A Simple Poverty Score for Peru. 2008, Grameen Foundation: St Louis, MO.
- [Background] Fernald LC, Kariger P, Hidrobo M, Gertler PJ. Socioeconomic gradients in child development in very young children: evidence from India, Indonesia, Peru, and Senegal. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17273-80. doi: 10.1073/pnas.1121241109. Epub 2012 Oct 8. PMID 23045688
- [Background] Rodriquez, S., ed. Escala de evaluacion del desarollo psicomotor: 0 a 24 meses. 12th ed ed. 1996, Galdoc: Santiago, Chile.
- [Background] Engle PL, Black MM, Behrman JR, Cabral de Mello M, Gertler PJ, Kapiriri L, Martorell R, Young ME; International Child Development Steering Group. Strategies to avoid the loss of developmental potential in more than 200 million children in the developing world. Lancet. 2007 Jan 20;369(9557):229-42. doi: 10.1016/S0140-6736(07)60112-3. PMID 17240290
- [Background] Lu C, Black MM, Richter LM. Risk of poor development in young children in low-income and middle-income countries: an estimation and analysis at the global, regional, and country level. Lancet Glob Health. 2016 Dec;4(12):e916-e922. doi: 10.1016/S2214-109X(16)30266-2. Epub 2016 Oct 4. PMID 27717632
- [Background] Becares L, Nazroo J, Kelly Y. A longitudinal examination of maternal, family, and area-level experiences of racism on children's socioemotional development: Patterns and possible explanations. Soc Sci Med. 2015 Oct;142:128-35. doi: 10.1016/j.socscimed.2015.08.025. Epub 2015 Aug 15. PMID 26301485
- [Background] Hanson JL, Chandra A, Wolfe BL, Pollak SD. Association between income and the hippocampus. PLoS One. 2011 May 4;6(5):e18712. doi: 10.1371/journal.pone.0018712. PMID 21573231
- [Background] Luby J, Belden A, Botteron K, Marrus N, Harms MP, Babb C, Nishino T, Barch D. The effects of poverty on childhood brain development: the mediating effect of caregiving and stressful life events. JAMA Pediatr. 2013 Dec;167(12):1135-42. doi: 10.1001/jamapediatrics.2013.3139. PMID 24165922
- [Background] Garner AS. Home visiting and the biology of toxic stress: opportunities to address early childhood adversity. Pediatrics. 2013 Nov;132 Suppl 2:S65-73. doi: 10.1542/peds.2013-1021D. PMID 24187125
- [Background] Grantham-McGregor SM, Powell CA, Walker SP, Himes JH. Nutritional supplementation, psychosocial stimulation, and mental development of stunted children: the Jamaican Study. Lancet. 1991 Jul 6;338(8758):1-5. doi: 10.1016/0140-6736(91)90001-6. PMID 1676083
- [Background] Munoz M, Nelson A, Johnson M, Godoy N, Serrano E, Chagua E, Valdivia J, Santacruz J, Wong M, Kolevic L, Kammerer B, Vega C, Vibbert M, Lundy S, Shin S. Community-Based Needs Assessment of Neurodevelopment, Caregiver, and Home Environment Factors in Young Children Affected by HIV in Lima, Peru. J Int Assoc Provid AIDS Care. 2017 Mar/Apr;16(2):161-167. doi: 10.1177/2325957416631625. Epub 2016 Jul 8. PMID 26917559
- See also: CASITA scale-up: Saving Brains Innovation — http://www.savingbrainsinnovation.net/projects/0769-05/